CLINICAL TRIAL: NCT05168891
Title: "Surgical Vs. Non-surgical Peri-implant Therapy: a 12-month Randomized Controlled Clinical Trial"
Brief Title: "Surgical Vs. Non-surgical Peri-implant Therapy"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Ramón Pons Calabuig, Dentistry, Master in Periodontics and Implants, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2019-05
Record Dates: First submitted 2021-11-11; First posted 2021-12-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2021-12

CONDITIONS: Peri-Implantitis; Implant Complication; Bone Loss
Keywords: peri-implantitis; non-surgical therapy; reconstructive therapy; bone graft
MeSH Terms: conditions — Peri-Implantitis; Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-blinded, randomized, controlled clinical trial with 1-year follow-up.
Who Masked: Investigator
Masking Description: Due to the nature of the study design, neither the patient nor the operator will be blinded. On the other hand, two blinded investigators will collect and record all the clinical and radiological measurements, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (TG) (Experimental): Patients will receive professional supragingival teeth/implant prophylaxis, oral hygiene instructions, and implant-supported prosthesis corrections if needed. After 1 week, peri-implant non-surgical therapy combined with antibiotic regimen consisting on metronidazole 500 mg every 8 hours for 7 days will be performed. Finally, the patients will be enrolled in a peri-implant maintenance therapy (PIMT) program every 3 months.
  Interventions: Procedure: Non-surgical therapy of peri-implantitis
- Control group (CG) (Experimental): Patients will receive professional supragingival teeth/implant prophylaxis, oral hygiene instructions, and implant-supported prosthesis corrections if needed. After 1 week, peri-implant non-surgical therapy combined with antibiotic regimen consisting on metronidazole 500 mg every 8 hours for 7 days will be performed. After one month, the regenerative surgical therapy will be performed as it follows: the intrabony component of the defect will be filled with a xenograft and covered with a collagen membrane allowing a non-submerged healing. Finally, the patients will be enrolled in a PIMT program every 3 months.
  Interventions: Procedure: Surgical therapy; Procedure: Non-surgical therapy of peri-implantitis

INTERVENTIONS:
Procedure: Surgical therapy — Peri-implantitis surgical therapy by means of open flap debridement, detoxification/decontamination of the implant surface and xenograft regeneration.
  Other Names: Reconstructive therapy for the management of peri-implantitis
  Arms: Control group (CG)
Procedure: Non-surgical therapy of peri-implantitis — Peri-implant non-surgical therapy combined with antibiotic regimen consisting on metronidazole 500 mg every 8 hours for 7 days will be performed
  Other Names: Non surgical debridement

SUMMARY:
The aim of this randomized clinical trial is to evaluate the effectiveness, in terms of clinical and radiographic changes, of non-surgical peri-implant therapy (mechanical/chemical) versus regenerative surgical therapy (xenograft and collagen membrane), after a follow-up period of 12 months.

DETAILED DESCRIPTION:
1. Objectives 1.1 Primary objective

   - To evaluate the radiographic bone fill of non-surgical mechanical debridement combined with systemic antibiotic therapy, compared to the adjunctive regenerative surgical therapy in the treatment of infraosseous peri-implant defects.

   1.2 Secondary objectives
   * To evaluate the following clinical parameters: modified plaque index (mPI), modified - Bleeding Index (mBI), BOP, SOP, implant PPD, mucosal recession (MR).
   * To evaluate the following radiographic outcomes: bone level (BL), intrabony defect (ID)
   * To evaluate the following Patient reported outcome measures (PROMs): Oral health impact profile (OHIP-14sp), VAS Score, pain medication.
2. Hypothesis

   - The non-surgical mechanical and antibiotic therapy of peri-implantitis in the treatment of infraosseous defects around implants will achieve similar radiographic bone fill and similar clinical results, when compared to the same protocol and the adjunction of a regenerative surgical therapy by means of xenograft plus a collagen membrane.
3. Material y methods:

3.1 Study design: This is a prospective, single-blinded, randomized, controlled clinical trial with 1-year follow-up.

3.2 Setting of the study Patients referred to Department of Periodontology (CUO) for treatment of periodontal and/or peri-implant diseases and who meet the inclusion criteria will be included in the study. Patients will be recruited consecutively. Furthermore, all study subjects will provide written informed consent before participating in the study. The present investigation will be performed following the principles outlined in the Declaration of Helsinki.

3.3 Study population To take part in this study, patients must present at least one implant diagnosed with peri-implantitis [i.e., peri-implant bone level ≥ 3mm apical to the most coronal portion of the intraosseous part of the implant, peri-implant pocket depth (PPD) ≥ 6 mm, and presence of bleeding and/or suppuration on gentle probing (BOP/SOP).

3.4 Randomization, allocation concealment and blindness The original participant identifiers (number of clinical history) will be replaced by new generated identifiers (code numbers) assigned according to patients' entrance in the study.

The randomization sequence will be carried out using a computer-generated list with a 1:1 allocation ratio according to a block randomization procedure (block size of four). Allocation concealment will be kept by means of opaque-sealed envelopes that will be opened immediately after the reevaluation of phase I therapy.

3.5 Sample size Using the radiographic bone fill as the primary outcome variable, the sample size has been calculated. Thirty-six patients (18 patients in each group) are necessary to detect a difference ≥ 0.5 mm in bone fill, assuming a common standard deviation of 0.41. This calculation assumes an alpha error of 0.05, a beta error of 0.1, and a statistical power of 90%. In addition, an estimation that 20% of subjects will be lost to follow-up has been taken into account.

3.6 Study visits 3.6.1 Screening examination Two calibrated investigators (C.V. and R.P.) will evaluate and enroll the patients. The clinicians will review with the patient the Information and Medication History Forms and record the information.

3.6.2 Treatment visits Baseline All subjects will receive a session of full-mouth professional prophylaxis, including scaling and tooth polishing. Supragingival debridement by means of an ultrasonic device using a plastic tip will be performed. Finally, the prosthetic components will be polished using a rubber cup.

Individualized instructions in proper oral hygiene measures will be given to all patients enrolled in the study.

Non-surgical therapy All the patients included in the study (both test and control groups) will received a peri-implant non-surgical therapy that will be standardized as follows: after local anesthesia (articaine 4% and adrenaline 1:100,000), the implant surfaces will be treated with ultrasonic devices with the H3 dental ultrasonic scaler. Curettage (SyG 7/89) of the bone defect will be performed and glycine air powder will be applied subgingivally (Air-flow®) with an air-flow piezon device.

After mechanical treatment, the antibiotic regimen consisting on metronidazole 500 mg every 8 hours for 7 days will be prescribed for all patients. Anti-inflammatory therapy was prescribed (ibuprofen 600 mg maximum thrice daily) for the first three days after the treatments. In addition, the use of additional pain killers (paracetamol every 4 hours) was recorded.

Six weeks after the non-surgical therapy, a clinical and radiographic evaluation will be performed. Immediately, an opaque-sealed envelope will be opened, and the patient will be assigned to test or control group.

Surgical therapy Patients assigned to the control group will undergo surgical peri-implant treatment that will be performed in the following way: after rinsing with 0.12% CHX for 1 minute and the appliance of local anesthesia, intrasulcular incisions will be designed and mucoperiosteal flaps will be raised. Granulation tissue will be removed using curettes and an ultrasonic device with the H3 dental ultrasonic. An implantoplasty procedure will be used to eliminate the supracrestal exposed moderate rough titanium surface of the implant using a diamond bur and surface will be polished with an Arkansas stone.

The infrabony component of the implant surface will be further decontaminated using ultrasonic scalers and with further chemical rinsing with 3% H2O2.

The intrabony component of the defect will be filled with a xenograft moistened in sterile saline for 5 minutes. Defects will be then covered with a collagen membrane over the entire defect. The flaps will be then repositioned with polypropylene 5/0 interrupted sutures allowing for a non-submerged healing.

Post-surgically, anti-inflammatory therapy will be prescribed for the first three days after the treatments and, according to the patients' individual needs, up to the first week. In addition, the use of additional pain killers will be recorded.

All patients will be recommended to use a 0.12% CHX mouth rinse, twice daily for 2 weeks. Finally, sutures will be removed after 15 days and patients will be reinstructed to re-install mechanical toothbrushing first with an ultra-soft brush for one week and then regular toothbrushing as explained during the initial therapy.

3.7.3 Follow-up visits Patients will be seen after 6 weeks from the non-surgical therapy, for the revaluation of the therapy and the first radiographic follow-up.

Patients of the control group will be seen after 6 weeks from the surgical therapy, for the revaluation of the therapy and the radiographic follow-up.

All patients (both test and control group) will be included in a peri-implant maintenance therapy (PIMT) program ever 3 months until the end of the study. At each PIMT visit, a clinical examination with the assessment of full mouth plaque index (FMPI) and full mouth bleeding index (FMBI), a reinforcement of oral hygiene instructions, supragingival and, if needed, subgingival debridement [BOP and/or peri-implant pocket depth (PPD) ≥ 5mm] as well as tooth polishing will be performed. Two of these visits will correspond to the radiographic examination and PROMs evaluation, at 6 and 12 months after the treatment.

3.8 Clinical and radiological examination 3.8.1 Demographic data An initial questionnaire will be conducted to obtain information regarding age, race, gender (female/male), medical history, medication, and health behavior (smoking habits). Smoking behavior will be specified as 3 categories: never smoker, former smoker, or current smoker (light smokers: < 10 cigarettes/day). Patients will be asked about their tobacco smoke exposure in terms of consumption (i.e. the number of cigarettes consumed per day); duration (i.e. the number of years of smoking); and lifetime exposure (i.e. the accumulated exposure as formed by the product of consumption and duration: cigarette-years). In case of former smokers, patients will be asked about the smoke-free time following cessation. Furthermore, implant position (maxilla/mandible and incisors, canines, premolars, and molars) and implant system will be further recorded as well as the type of prosthesis (cemented/screw-retained).

3.8.2 Clinical measurements

The following clinical parameters will be assessed for each implant by a single calibrated examiner (R.P.) at baseline and at 6 weeks, 6 and 12 months after the therapy using a periodontal probe:

1. Full mouth plaque index (FMPI) assessed dichotomously at four sites per tooth.
2. Full mouth bleeding index (FMBI) assessed dichotomously as presence or absence of bleeding after 30 seconds of gently probing.
3. Full mouth PD measured at six aspects around all teeth.
4. Modified plaque index (mPI) will be measured at six aspects around implants.
5. Modified bleeding index (mBI) will be assessed 30 seconds after 0.15 N force probing.

   This variable will be dichotomized in presence/absence of bleeding (BOP).
6. SOP evaluated after assessing dichotomously the presence of suppuration within 30 seconds after gentle probing.
7. Implant PPD, measured from the mucosal margin to the bottom of the probable pocket, determined at six aspects per implant: with a resin splint.
8. Mucosal recession (MR) at the implant will be recorded at six aspects per implant with a resin splint.

5.8.3 Radiographic examination A periapical radiograph will be obtained using the long-cone parallel technique and a film at baseline and six weeks, 6 and 12-month follow-up visit. All radiographs will be standardized in their exposure (7 mA-60 kV/20 ms).

The following measurements will be recorded by an independent previously calibrated examiner (M.C.S) at the mesial and distal aspects of the treated implants:

* Bone level (BL): distance (mm) between the implant shoulder and the base of the defect,
* Intrabony defect (ID), distance (mm) between the bottom of the defect and the line connecting the distal and mesial interproximal bone crest.

Radiographic bone fill (BF) will be calculated as it follows:

BF = (BLbaseline - BL6/12 months) / (IDbaseline) x 100 The measurements will be determined using an image-processing program (ImageJ)

5.8.4 Patient reported outcome measures (PROMs) Patients of test and control group will be subjected to the 14-items oral health-related quality of life (OHIP-14sp) questionnaire in the Spanish version at the baseline and after 6 weeks as well as 6 and 12 months of follow-up.

3.9 Intra-examiner reproducibility Reproducibility of radiographic and clinical examinations will be conducted by the repeated examination of radiographic bone level and PPD record of 5 implants in 5 patients, 1 week apart, before the beginning of the study.

3.10 Withdrawal of consent The Patient Information Sheet will clearly state that the patient can withdraw from the study at any time without prejudice or explanation. Such withdrawal will be documented in the medical record file. Losses to follow-up are taken into account in the sample size calculations (20%).

4. Statistical Analysis: The patient will be considered the unit of analysis. In order to describe the qualitative variables, absolute frequencies and percentages will be used. The description of quantitative variables will be performed using the mean, standard deviation (SD), median and quartiles. The Kolmogorov-Smirnov test will be used to assess the normality of distributions The results will be described with odds ratios (OR) with a 95% confidence interval (CI) and p-values. Level of significance will be set at 0.05. The SP

ELIGIBILITY:
To take part in this study, patients must present at least one implant diagnosed with peri-implantitis [i.e., peri-implant bone level ≥ 3mm apical to the most coronal portion of the intraosseous part of the implant, peri-implant pocket depth (PPD) ≥ 6 mm, and presence of bleeding and/or suppuration on gentle probing (BOP/SOP) (Berglunh et al. 2018)

Inclusion Criteria:

* Men and women over 18 years old.
* Presence of ≥ 1 endosseous implants with clinical and radiographic signs of peri- implantitis [i.e., peri-implant bone level ≥ 3mm apical to the most coronal portion of the intraosseous part of the implant, PPD ≥ 6 mm, and presence of bleeding and/or suppuration on gentle probing (BOP/SOP).
* Implant function time ≥ 1 year.
* Vertical peri-implant bone defect (defects of 2-3 walls and a defect depth ≥ 3 mm).
* Presence of at least 2 mm of keratinized mucosa.
* Absence of active periodontal disease.
* Good level of oral hygiene (Plaque Index < 25%) (O'Leary et al. 1972)
* Screw-retained single-unit crowns and partial dental prosthesis that allowed correct access for brushing; and, if not,
* Prostheses that could be modified.
* Absence of occlusal overload.

Exclusion Criteria:

* Clinical implant mobility.
* Radiographic peri-implant bone loss > 50%.
* Pregnancy or lactating females.
* Any medical condition which contraindicated surgical peri-implant therapy.
* Previous non-surgical treatment (i.e., subgingival debridement) of the affected implants at least 12 months before.
* Previous surgical treatment of the affected implants.
* Systemic diseases, medications, or conditions that may compromise wound healing influencing the outcome of the therapy.
* Known allergy or intolerance to metronidazole or ibuprofeno.
* Use of systemic antibiotics during the previous 3 months.
* Use of systemic antibiotics for endocarditis prophylaxis.
* Smoking more than 10 cigarettes/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Defect fil (mm) | 12 months after therapy
  peri-implant defect fill (≥1.0 mm and < 1 mm) from radiographic baseline

SECONDARY OUTCOMES:
Implant Pocket probing depth (PPD) (mm) | 12 months after therapy
  Measured from the mucosal margin to the bottom of the probable pocket, determined at six aspects per implant
modified Plaque Index (mPI) | 12 months after therapy
  measured at six aspects around implants and scored as: • Score 0 - no detection of plaque.
  * Score 1 - plaque only recognized by running a probe across the smooth marginal surface of the implant.
  * Score 2 - plaque can be seen by the naked eye.
  * Score 3 - abundance of soft matter.
modified Bleeding Index (mBI) | 12 months after therapy
  assessed 30 seconds after 0.15 N force probing and scored: • Score 0 - no bleeding.
  * Score 1 - isolated bleeding spots visible.
  * Score 2 - blood forms a confluent red line on margin.
  * Score 3 - heavy or profuse bleeding
Bleeding on probing (BOP) (%) | 12 months after therapy
  evaluated after assessing dichotomously the presence of bleeding within 30 seconds after gentle probing.
Suppuration on probing (SUP) (%) | 12 months after therapy
  evaluated after assessing dichotomously the presence of suppuration within 30 seconds after gentle probing.
Bone level (BL) changes | 12 months after therapy
  Distance (mm) between the implant shoulder and the base of the defect.
Intrabony defect (ID) changes | 12 months after therapy
  distance (mm) between the bottom of the defect and the line connecting the distal and mesial interproximal bone crest
Oral health impact profile (OHIP-14sp) | 12 months after therapy
  Patient reported outcome measures (PROMS) by means of a questionnaire
VAS Score | 12 months after therapy
  after non-surgical therapy and surgical therapy pain will be assessed using a visual analogue scale (VAS score; VAS 0-100, 100 reflecting the highest morbidity).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, PhD, Study Chair — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya (UIC), Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No